CLINICAL TRIAL: NCT06905509
Title: A Phase 2 Study of Epcoritamab (Epco) Plus Physician's Choice of Platinum-Containing Chemotherapy Pre-Autologous Hematopoietic Cell Transplantation (AutoHCT) Followed by Post-AutoHCT Epco Consolidation/ Maintenance in Relapsed/ Refractory Large B-Cell Lymphoma (R/R LBCL)
Brief Title: Epcoritamab Plus Standard of Care Platinum-Based Chemotherapy and Autologous Hematopoietic Cell Transplant for the Treatment of Relapsed or Refractory Large B-cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Joseph Tuscano (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Joseph Tuscano, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC316; NCI-2025-01557 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCDCC316 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH)
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Recurrent High Grade B-Cell Lymphoma With MYC and BCL2 Rearrangements; Recurrent High Grade B-Cell Lymphoma With MYC and BCL6 Rearrangements; Recurrent High Grade B-Cell Lymphoma, Not Otherwise Specified; Recurrent Nodal Marginal Zone Lymphoma; Recurrent Transformed Follicular Lymphoma to Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Refractory High Grade B-Cell Lymphoma With MYC and BCL2 Rearrangements; Refractory High Grade B-Cell Lymphoma With MYC and BCL6 Rearrangements; Refractory High Grade B-Cell Lymphoma, Not Otherwise Specified; Refractory Nodal Marginal Zone Lymphoma; Refractory Transformed Follicular Lymphoma to Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, B-Cell, Marginal Zone | interventions — Stem Cell Transplantation; Carboplatin; Cytarabine; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; etoposide phosphate; Gemcitabine; Ifosfamide; Oxaliplatin; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (epcoritamab, SOC chemotherapy, autoHCT) (Experimental): See Detailed Description
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Carboplatin; Drug: Cytarabine; Drug: Dexamethasone; Biological: Epcoritamab; Drug: Etoposide Phosphate; Drug: Gemcitabine; Drug: Ifosfamide; Procedure: Multigated Acquisition Scan; Drug: Oxaliplatin; Biological: Rituximab

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo autoHCT
  Other Names: AHSCT; Autologous; Autologous Hematopoietic Cell Transplantation; Autologous Stem Cell Transplant; Autologous Stem Cell Transplantation; Stem Cell Transplantation, Autologous
Drug: Carboplatin — Given carboplatin
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cytarabine — Given cytarabine
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Dexamethasone — Given dexamethasone
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; LenaDex; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Biological: Epcoritamab — Given SC
  Other Names: Anti-CD20/CD3 Bispecific Antibody GEN3013; DuoBody-CD3xCD20; Epcoritamab-bysp; Epkinly; GEN 3013; GEN-3013; GEN3013; Tepkinly
Drug: Etoposide Phosphate — Given etoposide phosphate
  Other Names: Etopophos
Drug: Gemcitabine — Given gemcitabine
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
Drug: Ifosfamide — Given ifosfamide
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Oxaliplatin — Given oxaliplatin
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; Elplat; JM 83; JM-83; JM83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; RP54780; SR 96669; SR-96669; SR96669
Biological: Rituximab — Given rituximab
  Other Names: ABP 798; ABP-798; ABP798; BI 695500; BI-695500; BI695500; Blitzima; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT P10; CT-P10; CTP10; GP 2013; GP-2013; GP2013; IDEC 102; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; IDEC102; Ikgdar; Mabtas; MabThera; Monoclonal Antibody IDEC-C2B8; PF 05280586; PF-05280586; PF05280586; Riabni; Ritemvia; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar GP2013; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; Rituximab-abbs; Rituximab-arrx; Rituximab-blit; Rituximab-pvvr; Rituximab-rite; Rituximab-rixa; Rituximab-rixi; Rixathon; Riximyo; RTXM 83; RTXM-83; RTXM83; Ruxience; Truxima

SUMMARY:
This phase II trial tests how well epcoritamab in combination with standard of care (SOC) platinum-based chemotherapy (rituximab, ifosfamide, carboplatin, etoposide [RICE], rituximab, cytarabine, dexamethasone, oxaliplatin or carboplatin RDHAP/X] or gemcitabine and oxaliplatin [Gem/Ox]) and autologous hematopoietic cell transplant (HCT) works in treating patients with large B-cell lymphoma (LBCL) that has come back after a period of improvement (relapsed) or that has not responded to previous treatment (refractory). Epcoritamab, a type of bispecific T-cell engager, binds to a protein called CD3, which is found on T cells (a type of white blood cell). It also binds to a protein called CD20, which is found on B cells (another type of white blood cell) and some lymphoma cells. This may help the immune system kill cancer cells. Carboplatin is in a class of medications known as platinum-containing compounds. It works in a way similar to the anticancer drug cisplatin, but may be better tolerated than cisplatin. Carboplatin works by killing, stopping or slowing the growth of cancer cells. Oxaliplatin is in a class of medications called platinum-containing antineoplastic agents. It damages the cell's deoxyribonucleic acid (DNA) and may kill cancer cells. Rituximab is a monoclonal antibody. It binds to a protein called CD20, which is found on B cells and some types of cancer cells. This may help the immune system kill cancer cells. Chemotherapy drugs, such as ifosfamide, etoposide phosphate, cytarabine, and gemcitabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Dexamethasone is in a class of medications called corticosteroids. It is used to reduce inflammation and lower the body's immune response to help lessen the side effects of chemotherapy drugs. An autologous HCT is a procedure in which blood-forming stem cells (cells from which all blood cells develop) are removed, stored, and later given back to the same person. Giving epcoritamab in combination with SOC platinum-based chemotherapy, such as RICE, RDHAP/X and Gem/Ox, and autologous HCT may kill more cancer cells in patients with relapsed or refractory LBCL.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the anti-tumor activity of epcoritamab + platinum-containing chemotherapy + autologous HCT therapy in patients with relapsed or refractory (R/R) LBCL.

SECONDARY OBJECTIVES:

I. To evaluate the toxicities of epcoritamab + platinum-containing chemotherapy with or without autologous HCT therapy in patients with R/R LBCL.

II. To further assess the anti-tumor activity of epcoritamab + platinum-containing chemotherapy + autologous HCT therapy in patients with R/R LBCL.

OUTLINE:

PRE-AUTOHCT: Patients receive epcoritamab subcutaneously (SC) on days 1, 8, 15, and 22 of each cycle. Cycles repeat every 28 days for up to 3 cycles without disease progression or unacceptable toxicity. Patients may also receive rituximab, cytarabine, dexamethasone, oxaliplatin, or carboplatin once every 21 days for cycles 1-3 or gemcitabine and oxaliplatin once every 2 weeks of each 28-day cycle for cycles 1-3 or rituximab, ifosfamide, carboplatin and etoposide phosphate once every 21 days of cycles 1-3 per SOC.

AUTOHCT: Patients undergo autoHCT on week 0 per SOC.

POST-AUTOHCT/CONSOLIDATION: Patients receive epcoritamab SC on days 1, 8, 15, and 22 of cycles 1-3, on days 1 and 15 of cycles 4-9, and on day 1 of the remaining cycles. Cycles repeat every 28 days for up to 12 cycles without disease progression or unacceptable toxicity.

Patients also undergo echocardiography (ECHO) or multigated acquisition scan (MUGA) at screening and as clinically indicated, and blood sample collection and computed tomography (CT) or positron emission tomography (PET)/CT throughout the study. Additionally, patients may undergo brain magnetic resonance imaging (MRI) or CT at screening.

After completion of study treatment, patients are followed up at 30 days then every 4 months for up to 2 years post autoHCT.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed R/R LBCL

  * Can include diffuse large B-cell lymphoma (DLBCL) (not otherwise specified [NOS] or with concurrent MYC and BCL2 rearrangements), high-grade B-cell lymphoma (HGBCL) (NOS or with MYC and BCL2 or BCL6 rearrangements) and transformed follicular lymphoma (FL) and nodal marginal zone lymphoma (MZL)
  * Histological confirmed CD20+ relapsed/ refractory large cell lymphoma
* Must have had relapsed or refractory disease following standard frontline chemotherapy. Refractory disease is defined as large cell lymphoma not achieving complete remission, progressing, or relapsing within 6 months after first-line chemotherapy based on PET/CT per the Lugano criteria. Relapsed disease is defined as disease that recurs beyond 6 months after completion of initial chemotherapy based on PET/CT per the Lugano criteria
* Have received 1 or more prior lines of systemic therapy for the treatment of large cell lymphoma. NOTE: Prior radiation therapy or systemic corticosteroids will not be considered a line of therapy
* Candidate for platinum-containing chemotherapy (RICE, RDHAP/X, or R-Gem/Ox) pre-autologous hematopoietic cell transplantation (autoHCT) followed by autoHCT as per institutional guidelines
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%)
* Measurable disease via diagnostic quality CT or PET/CT with at least 1 node having the longest diameter (LDi) greater than (>) 1.5 centimeter (cm) or 1 extranodal lesion with LDi > 1 cm (per the Lugano criteria 2014)
* Aged ≥ 18 at the time of consent
* Creatinine clearance (CrCl) ≥ 45 mL/min (Cockcroft-Gault)
* Serum alanine aminotransferase (ALT) ≤ 3 x upper limit of normal (ULN)
* Serum aspartate aminotransferase (AST) ≤ 3 x ULN
* Bilirubin ≤ 1.5 x ULN unless due to Gilbert's syndrome or controlled autoimmune hemolytic anemia (not requiring immunosuppressive other than ≤ 20 mg of prednisolone daily)

  * Note: Patients with Gilbert's syndrome may be included if total bilirubin is ≤ 3 x ULN and direct bilirubin is ≤ 1.5 x ULN
* Hemoglobin ≥ 8.0 g/dL

  * Note: Blood transfusion may be administered during Screening to meet this requirement only if anemia is due to marrow involvement of non-Hodgkin lymphoma (NHL)
* Absolute neutrophil count ≥ 1000/uL

  * Note: Growth factor support is allowed to meet this requirement at Screening only if directly attributable to NHL infiltration of the bone marrow, proven by bone marrow biopsy
* Platelet count ≥ 75,000/uL or ≥ 50,000/uL if bone marrow (BM) involvement or splenomegaly

  * Note: Transfusion may be administered during screening to meet this requirement
* prothrombin time (PT)/international normalized ratio (INR)/activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN
* Note: If any of the above-mentioned cytopenias are present, there should be no evidence of myelodysplastic syndrome (MDS) or hypoplastic bone marrow
* HIV-infected patients on effective anti-retroviral therapy with stable viral load and CD4 count for 1 year prior to enrollment are eligible for this trial. Testing for HIV viral load and antibody at screening is mandatory
* Patients with a history of chronic hepatitis B virus (HBV) infection, must have an undetectable HBV viral load on suppressive therapy, if indicated. Patients with evidence of prior HBV but who are polymerase chain reaction (PCR)-negative are permitted in the trial but should receive prophylactic antiviral therapy. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, the HCV viral load must be undetectable to be eligible for this trial. Patients who received treatment for HCV that was intended to eradicate the virus may participate if hepatitis C ribonucleic acid (RNA) levels are undetectable. Testing for HBV and HCV is mandatory at screening
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 12 months after the last dose of epcoritamab
* Provision of signed and dated informed consent form

Exclusion Criteria:

* Any adverse event (AE) related to the previous large cell lymphoma therapy which has not recovered to grade ≤ 1 (Common Terminology Criteria for Adverse Events [CTCAE] version [v.] 5.0) or baseline by cycle 1 day 1 (C1D1), except alopecia and non-clinically significant laboratory abnormalities
* Uncontrolled intercurrent illness (including infection)
* Known active central nervous system or meningeal (including leptomeningeal) involvement. Patients diagnosed with central nervous system (CNS) disease who achieved and maintained CNS complete response (CR) at the time of relapse are eligible. Lumbar puncture must be done in this case prior to study entry (within 90 days of enrollment) to demonstrate CNS CR status. Tests to investigate CNS involvement are required otherwise only if clinically indicated (i.e. disease suspected on basis of symptoms or other findings)
* Receiving any other investigational treatments
* Previous treatment with any bispecific T-cell engager with or without chemotherapy
* Treatment with an investigational drug within 4 weeks or 5 half-lives, whichever is longer, prior to the first dose of epcoritamab
* Concurrent use of other anti-cancer agents or treatments except for certain therapeutics (e.g., prostate, breast hormonal-based therapy) per the treating physician's discretion

  * Standard agents within 2 weeks or 5 half-lives, whichever is shorter, prior to the first dose of epcoritamab (excluding anti-CD20 monoclonal antibodies [mAbs], which can be administered until first full dose of epcoritamab); or
  * CAR-T cell therapy within 30 days prior to the first dose of epcoritamab
  * Palliative radiation is permitted only if on non-target lesions
* Motor and sensory neuropathy grade ≥ 2 (CTCAE v.5.0)
* Patients with a history of other malignancies, except adequately treated non-melanoma skin cancer, non-invasive superficial bladder cancer, curatively treated in-situ cancer of the cervix, ductal carcinoma in situ (DCIS) of the breast, localized low grade prostate cancer (up to Gleason score 6), or other solid tumors curatively treated with no evidence of disease for at least 3 years
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at trial enrollment or significant infections within 2 weeks prior to the first dose of epcoritamab
* Confirmed history or current autoimmune disease or other diseases requiring permanent immunosuppressive therapy. Low-dose (10 mg/day) prednisolone (or equivalent) for rheumatoid arthritis or similar conditions is allowed
* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study)
* Participant received any prior allogeneic hematopoietic stem cell transplantation (HSCT) or solid organ transplantation
* Autoimmune disease or other diseases that require continuous immunosuppressive therapy (except for prednisone doses of less than or equal to 10 mg, which is allowed)
* Uncontrolled autoimmune hemolytic anemia or immune thrombocytopenia (requiring > 20 mg of prednisolone daily) or other concurrent uncontrolled medical conditions
* Clinically significant cardiac disease including but not limited to:

  * Unstable or uncontrolled disease/condition related to or affecting cardiac function, e.g., unstable angina, congestive heart failure grade III or IV as classified by the New York Heart Association, uncontrolled clinically significant cardiac arrhythmia (CTCAE v 5.0 grade 2 or higher), or clinically significant electrocardiogram (ECG) abnormalities. Controlled New York Heart Association (NYHA) grade 1 or 2 are eligible
  * Myocardial infarction, intracranial bleed, or stroke within the past 6 months
  * Screening 12-lead ECG showing a baseline QT interval as corrected by Fridericia's formula (QTcF) > 480 msec. NOTE: This criterion does not apply to participants with a left bundle branch block
  * In case of any history of cardiovascular disease, a cardiology consult is required within 60 days prior to enrollment
  * Age ≥ 75 and 2 or more active grade ≥ 2 cardiovascular conditions
* Prior treatment with live, attenuated vaccines within 28 days prior to initiation of epcoritamab. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, bacillus Calmette-Guerin, and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed. Food and Drug Administration (FDA)-approved severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) vaccinations allowed
* Immune effector cell encephalopathy (ICE) score of less than 10 at study entry
* Suspected allergies, hypersensitivity, or intolerance to epcoritamab or another anti-CD20 mAb or its excipients
* Active HBV (DNA PCR-positive). Patients with evidence of prior HBV but who are PCR-negative are permitted in the trial but should receive prophylactic antiviral therapy
* Active hepatitis C (RNA PCR-positive infection). Patients who received treatment for HCV that was intended to eradicate the virus may participate if hepatitis C RNA levels are undetectable
* Known history of seropositivity for HIV infection
* Active cytomegalovirus (CMV) infection (PCR positive)
* Pregnant, breastfeeding, or planning to become pregnant while enrolled in this trial or within 12 months after the last dose of epcoritamab
* Plans to donate sperm or conceive a child through intercourse while enrolled in this trial or within 12 months after the last dose of epcoritamab
* Ongoing active bacterial, viral, fungal, mycobacterial, parasitic, or other infection requiring systemic treatment (excluding prophylactic treatment) at the time of enrollment or within the previous 2 weeks prior to the first dose of epcoritamab
* Known active severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection. If a subject has signs/symptoms suggestive of SARS-CoV-2 infection or have had recent known exposure to someone with SARS-CoV-2 infection, the subject must have a negative molecular (e.g., PCR) test, or 2 negative antigen test results at least 24 hours apart, to rule out SARS-CoV-2 infection. Note: SARS-CoV-2 diagnostic tests should be applied following local requirements/recommendations. Subjects who do not meet SARS-CoV-2 infection eligibility criteria must be screen failed and may only rescreen per criteria
* Suspected active or inadequately treated latent tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
Complete response rate (CRR) | From first dose up to 2 years post-autologous hematopoietic cell transplantation (autoHCT) therapy
  Will be assessed by Lugano 2014. Will be calculated as the number of participants achieving complete response divided by the number of evaluable patients. CRR will be presented alongside the corresponding exact binomial 95% confidence interval.

SECONDARY OUTCOMES:
Incidence of treatment-related adverse events (AEs) | From first dose through 30 days post last epcoritamab dose
  The proportion of participants experiencing AEs, serious AEs, and treatment delays will be summarized. All AEs will be listed, documenting the course, outcome, severity, and relationship to the study treatment. Incidence rates of AEs and the proportion of participants prematurely withdrawn from the study due to AEs will be reported. Will be classified by severity, and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
Progression-free survival | From the date of enrollment until the first occurrence of disease progression, or death from any cause, whichever occurs first, assessed up to 2 years post-autoHCT therapy
  Will be summarized using the Kaplan-Meier method. Summary statistics will include median and event-free probabilities at pre-specified time points, along with their associated two-sided 95% confidence intervals (CIs).
Objective response | From first dose up to 2 years post-autoHCT therapy
  Will be assessed by Lugano 2014. Will be presented using descriptive statistics. Tabulations will be produced for appropriate disposition, demographic, baseline, and efficacy parameters. For continuous variables, the number of participants, mean, median, standard deviation, minimum, and maximum values will be presented. For categorical variables, numbers and percentages of participants within each category (with a category for missing data) will be presented along with binomial exact 95% CIs, unless stated otherwise.
Overall survival | From first dose to death due to any causes, assessed up to 2 years post-autoHCT therapy
  Will be summarized using the Kaplan-Meier method. Summary statistics will include median and event-free probabilities at pre-specified time points, along with their associated two-sided 95% confidence intervals.
Duration of minimal residual disease (MRD) negativity | Pre-autoHCT and 90 days post-autoHCT
  Will be presented using descriptive statistics. Tabulations will be produced for appropriate disposition, demographic, baseline, and efficacy parameters. For continuous variables, the number of participants, mean, median, standard deviation, minimum, and maximum values will be presented. For categorical variables, numbers and percentages of participants within each category (with a category for missing data) will be presented along with binomial exact 95% CIs, unless stated otherwise. Will be calculated by dividing the number of participants with at least one MRD-negative result within 3 cycles of consolidation therapy by the total number of participants who undergo circulating tumor derived deoxyribonucleic acid (ctDNA) MRD testing.
MRD negativity | Pre-autoHCT and 90 days post-autoHCT
  Will be presented using descriptive statistics. Tabulations will be produced for appropriate disposition, demographic, baseline, and efficacy parameters. For continuous variables, the number of participants, mean, median, standard deviation, minimum, and maximum values will be presented. For categorical variables, numbers and percentages of participants within each category (with a category for missing data) will be presented along with binomial exact 95% CIs, unless stated otherwise. Will be calculated by dividing the number of participants with at least one MRD-negative result within 3 cycles of consolidation therapy by the total number of participants who undergo ctDNA MRD testing.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Tuscano, Study Chair — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States